CLINICAL TRIAL: NCT04260555
Title: A Multicenter, Randomized, Double-Blind, Parallel, Active-controlled, Superiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW1601 Compared to DW16011 and DW16012 for Acute Bronchitis
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of 'DW1601' in Acute Bronchitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1601-301
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEST (Experimental): tid PO, DW1601 20ml + Placebo of DW16011 20ml + Placebo of DW16012 9ml
  Interventions: Drug: DW1601
- Reference 1 (Active Comparator): tid PO, Placebo of DW1601 20ml + DW16011 20ml + Placebo of DW16012 9ml
  Interventions: Drug: DW16011
- Reference 2 (Active Comparator): tid PO, Placebo of DW1601 20ml + Placebo of DW16011 20ml + DW16012 9ml
  Interventions: Drug: DW16012

INTERVENTIONS:
Drug: DW1601 — Total 7 days of treatment and The daily dose is tid. (DW1601 20ml + Placebo of DW16011 20ml + Placebo of DW16012 9ml)
  Arms: TEST
Drug: DW16011 — Total 7 days of treatment and The daily dose is tid. (Placebo of DW1601 20ml + DW16011 20ml + Placebo of DW16012 9ml)
  Arms: Reference 1
Drug: DW16012 — Total 7 days of treatment and The daily dose is tid. (Placebo of DW1601 20ml + Placebo of DW16011 20ml + DW16012 9ml)
  Arms: Reference 2

SUMMARY:
A Multicenter, Randomized, Double-Blind, Parallel, Active-controlled, Superiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW1601 Compared to DW16011 and DW16012 for Acute Bronchitis

ELIGIBILITY:
Inclusion Criteria:

* Both gender, 19 years ≤ age ≤ 80 years
* Bronchitis Severity Score* ≥ 5point at Visit 2 (Randomized Visit)
* Acute bronchitis within 48hr based on Visit 2 (Randomized Visit)
* Those who can comply with the requirements of clinical trials
* Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

* Patients who investigators determines to severe respiratory disease that would interfere with study assessment
* Patients with systemic infections requiring systemic antibiotic therapy
* patient with hemostatic disorder

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Bronchitis Severity Score(BSS) | Day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea